CLINICAL TRIAL: NCT02079948
Title: Role of Methotrexate in Improving Physical Function in Older Adults With Elevated Levels of Inflammation
Brief Title: Inflammation Control For Elders: ICE Study
Acronym: ICE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Potential participants had concerns about taking the study drug (methotrexate).
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1182013; P30AG028740 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Inflammation; Aging
Keywords: Aging; Cognitive Function; Physical Function; Systematic Inflammation; Methotrexate; Pain Symptoms
MeSH Terms: conditions — Inflammation; Pain | interventions — Methotrexate; Folic Acid; microcrystalline cellulose; Magnetic Resonance Spectroscopy; X-Rays; Biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Methotrexate + Folic Acid (Active Comparator): Participants in the methotrexate condition will consume a dose of 15 mg/week of methotrexate during months 2 - 6. Participants will also consume 1 mg of folic acid/day for six days per week.
  Interventions: Procedure: Functional MRI Experimental Tasks; Procedure: Muscle Biopsy
- Placebo + Folic Acid (Placebo Comparator): Participants in the placebo condition will consume microcrystalline cellulose once per week. The number of capsules consumed on this day will match the number of capsules consumed by participants in the methotrexate condition. There are no active ingredients in the placebo capsules.
  Interventions: Procedure: Functional MRI Experimental Tasks; Procedure: Muscle Biopsy
- Functional MRI Experimental Tasks (Experimental): 15 participants will be randomly assigned to complete the fMRI visits at the baseline and 6 month.
  Interventions: Drug: Methotrexate + Folic Acid; Drug: Placebo + Folic Acid
- Muscle Biopsy (Experimental): 10 participants will be randomly assigned to complete the skeletal muscle tissue sample at the baseline and 6 month visits.
  Interventions: Drug: Methotrexate + Folic Acid; Drug: Placebo + Folic Acid

INTERVENTIONS:
Drug: Methotrexate + Folic Acid — Participants in the methotrexate + folic acid condition will have a
  * Blood draw at each monthly visit
  * Cognitive performance testing to assess memory performance
  * Physical function testing to assess walking speed and measure muscle endurance
  * Pain assessment testing to assess the presence and location of daily pain
  * Self-reported function and quality of life to measure disability and mobility limitations, and
  * Depression assessment testing to assess participants' level of depression.
  Other Names: Trexall; Rheumatrex
  Arms: Functional MRI Experimental Tasks; Muscle Biopsy
Drug: Placebo + Folic Acid — Participants in the placebo + folic acid condition will have a
  * Blood draw at each monthly visit
  * Cognitive performance testing to assess memory performance
  * Physical function testing to assess walking speed and measure muscle endurance
  * Pain assessment testing to assess the presence and location of daily pain
  * Self-reported function and quality of life to measure disability and mobility limitations, and
  * Depression assessment testing to assess participants' level of depression
  Other Names: Microcrystalline Cellulose
  Arms: Functional MRI Experimental Tasks; Muscle Biopsy
Procedure: Functional MRI Experimental Tasks — Participants who are randomly assigned to the fMRI scan wil receive their study drugs at the the Baseline fMRI visit. Participants who are randomly assigned to the fMRI will also attend complete their last visit at the 6 month period.
  Other Names: - MRI; -Magnetic Resonance (MR); -Nuclear Magnetic Resonance (NMR) Imaging
  Arms: Methotrexate + Folic Acid; Placebo + Folic Acid
Procedure: Muscle Biopsy — Participants who are randomly assigned to the muscle biopsy assessment of the study will receive their study drugs at the Baseline muscle biopsy visit. Participants who are randomly assigned to the muscle biopsy portion of the study will also complete their last visit at the 6 month period.
  Other Names: -Biopsy; -Muscle Tissue Sample
  Arms: Methotrexate + Folic Acid; Placebo + Folic Acid

SUMMARY:
This study will be the first to test whether a selected anti-inflammatory agent, methotrexate, reduces inflammation in a human body, improve cognitive and physical function, and reduce pain levels in older adults at risk for functional decline, due to systemic inflammation.

DETAILED DESCRIPTION:
If you decide to take part in this study, you will be randomly assigned (much like the flip of a coin) to receive either methotrexate or placebo. A placebo is a substance that looks like and is given in the same way as an experimental treatment but contains no medicine, for example [a sugar pill, an injection of saline (salt water)]. A placebo is used in research studies to show what effect a treatment has compared with taking nothing at all. If you are assigned to receive placebo, you will not receive the benefits of the methotrexate, if there are any, nor will you be exposed to its risks, which are described below under "What are the possible discomforts and risks?" Studies have shown, however, that about 1 in 3 persons who take a placebo do improve, if only for a short time. You and the physician and other persons doing the study will not know whether you are receiving placebo or methotrexate, but that information is available if it is needed. Also, you will have a 50% chance of receiving methotrexate and a 50% chance of receiving placebo.

Methotrexate lowers folate (vitamin B9) levels in the body, so when someone takes methotrexate, he/she needs to take folic acid. To make sure that methotrexate lowers levels of inflammation in the body and not folate, study participants in both groups will be given folic acid.

In the remainder of the description of what will be done, both the methotrexate and the placebo will be called "study treatment."

You will be given a study letter that describes the study. You will be asked to show this letter to your doctors and other medical specialists, so they know that you are participating in a study with study drugs.

You will be asked to take your study drugs every morning by mouth on an EMPTY STOMACH before breakfast. The study capsules containing methotrexate and the placebo will look the same.

Participants in the methotrexate group will slowly increase the amount of methotrexate they take in the first month up to the 15 mg/week. In the first week, participants will take 5 mg/week (i.e., 1 capsule on Day 7), in the second and third week they will take 10 mg/week (i.e., 2 capsules on Day 7), and in the fourth week they will take 15 mg/week (i.e., 3 capsules on Day 7). On Days 1-6, participants will take 1 folic acid capsule.

Participants in the placebo group will slowly increase the number of placebo capsules they take in the first month. In the first week, participants will take 1 placebo capsule on Day 7, in the second and third week they will take 2 placebo capsules on Day 7, and in the fourth week they will take 3 placebo capsules on Day 7. On Days 1-6, participants will take 1 folic acid capsule.

Store study medications at room temperature between 59° to 86°F (15° to 30°C) and keep them away from light.

Keep these and all medicines out of the reach of children.

You will be asked to take the study drugs for 6 months, and your participation in the study will last approximately 8 months. The investigators will ask you to attend 12 study visits at the research center located at the Institute on Aging - Clinical & Translational Research Building (IOA - CTRB):

1. Screening Visit
2. Baseline Visit
3. Baseline Functional Magnetic Imaging (fMRI) Visit
4. 1-Month Visit
5. 2-Month Visit
6. 3-Month Visit
7. 4-Month Visit
8. 5-Month Visit
9. 6-Month Visit
10. 6-Month fMRI Visit
11. Follow-Up Visit I
12. Follow-Up Visit II

The investigators will also call you approximately 9 times during the study to ask you how you feel and to find out if you remembered to take all your study drugs.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or over
* Blood Level of IL-6: > 2.54 pg/mL
* Physical Activity: < 120 minutes of moderate intensity physical activity per week
* Mild-to-moderate physical impairment: (SPPB < 9)
* Blood Pressure: < 160/90 mm Hg
* Willing and able to give informed consent

Exclusion Criteria:

* Significant underlying disease that is likely to limit participation and/or increase risk of interventions
* History or diagnosis of cardiovascular disease, myocardial infarction (heart attack), cerebrovascular accident, or unstable angina NYHA Class 3 or 4 congestive heart failure; aortic stenosis; cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina within the past 6 months;
* History or diagnosis of severe lung disease within the past 6 months
* Known chronic pericardial effusion, pleural effusion, or ascites; chronic liver disease; myeloproliferative disorders in the past 5 years; Lymphoproliferative disease diagnosed and/or treated within the last five years; non-basal cell malignancy
* Prior history of chronic infectious disease, renal insufficiency, interstitial lung disease, pneumonitis, bronchiectasis, pulmonary fibrosis, or pulmonary disease
* Cognitive impairment and/or diagnosis of dementia
* Failure to provide informed consent
* Current usage of methotrexate therapy
* Consume alcohol and refuses to reduce alcohol use to 3 or fewer drinks per week during the study
* History of drug or alcohol abuse or excessive alcohol use within past six months
* Abnormal laboratory values
* White blood cell count < 4,000/ul, hematocrit < 32%, or platelet count < 75,000/ul
* Liver transaminase levels (AST or ALT) > upper limit of normal (ULN) or albumin < the lower limit of normal (LLN)
* Creatinine clearance < 40 ml/min as estimated with the Cockroft-Gault equation
* Hypercalcemia (calcium > 10.4 mg/dL), hypocalcemia (calcium < 8.6 mg/dL), renal insufficiency (estimated glomerular filtration rate (eGFR) < 50 ml/min)
* Lives in a nursing home
* Self-reported inability to walk one block without any type of assistive device
* Chest pain or severe shortness of breath during the 400-meter walk test
* Terminal illness with life expectancy less than 12 months, as determined by a physician
* Medication exclusions (current use of anabolic medications [i.e., growth hormones or testosterone], antipsychotic agents, monoamine oxidase inhibitors, anticholinesterase inhibitors [i.e., Aricept], anticoagulant therapies [aspirin use is permitted], antibiotics for HIV or TB, or antibiotics for other uses currently or within the past two months)
* Chronic use of oral steroid therapy or other immunosuppressive or biologic response modifiers
* Requirement for use of drugs that alter folate metabolism or reduce tubular excretion or known allergies to antibiotics making avoidance of trimethoprim impossible
* Planning to leave the area in the next year
* Current smoker or less than 3 years quit
* Men who plan to father children during the study period or who are unwilling to use effective forms of contraception
* Women of child bearing potential
* Other significant co-morbid disease (e.g., renal failure on hemodialysis)
* Contraindications to fMRI (ex. cardiac pacemaker)
* Participating in another clinical trial or has received an investigational product within 30 days prior to screening/enrollment
* Any other condition that in the opinion of the principal investigator may compromise the participation in the study
* Participants with contraindications to the muscle biopsy procedure can participate in the study but will not be asked to participate in the muscle biopsy procedure.

The temporary exclusions include the following:

* Recent bacterial/viral infection (< 2 weeks)
* Acute febrile illness in prior 2 months
* Major surgery or hip/knee replacement in the past 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Markers of Systemic Inflammation | 6 Months
  To examine the effects of methotrexate on changes in markers of systemic inflammation (e.g., IL-6, CRP) and cellular inflammation (e.g., IL-6, TNF-α, and IL11β).

SECONDARY OUTCOMES:
Physical Function | 6 Months
  To examine the effects of methotrexate on changes in physical function (walking speed, muscle fatigue, and strength).
Cognitive Performance | 6 Months
  To examine the effects of methotrexate on cognitive performance (attention and memory).
Pain Symptoms | 6 Months
  To examine the effects of methotrexate on pain symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anton, PhD, Principal Investigator — University of Florida, Institute on Aging